CLINICAL TRIAL: NCT04818762
Title: Peripheral Fractional Tissue Oxygen Extraction and Infection in Term and Preterm Neonates - a Prospective Pilot Observational Study
Brief Title: Peripheral Fractional Tissue Oxygen Extraction and Infection in Term and Preterm Neonates
Acronym: pFTOE
Status: Recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: pFTOE
Record Dates: First submitted 2021-03-15; First posted 2021-03-26 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Neonatal Infection; Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Preterm neonates with infection: Preterm neonates (30+0 - 36+6 weeks of gestation) with clinical and laboratory signs of early onset infection (within 72 hours after birth).
- Preterm neonates without infection: Preterm neonates (30+0 - 36+6 weeks of gestation) without clinical and laboratory signs of early onset infection (within 72 hours after birth).
- Term neonates with infection: Preterm neonates (30+0 - 36+6 weeks of gestation) with clinical and laboratory signs of early onset infection (within 72 hours after birth).
- Term neonates without infection: Preterm neonates (30+0 - 36+6 weeks of gestation) without clinical and laboratory signs of early onset infection (within 72 hours after birth).

SUMMARY:
This is a prospective observational pilot study investigating if peripheral fractional tissue oxygen extraction (pFTOE) measured by five short near-infrared spectroscopy (NIRS) (re-)applications within the first 6 hours after birth in neonates with respiratory distress differs in neonates with early onset infection and neonate without infection

DETAILED DESCRIPTION:
Background Near-infrared spectroscopy (NIRS) enables non-invasive, continuous monitoring of oxygenation and perfusion in different tissues. In several studies NIRS has been described to have the potential to detect centralisation due to perfusion heterogeneity, arterio-venous shunting and impaired autoregulation. Thus, peripheral muscle NIRS measurement has the potential to provide information at early stages of inflammation also due to infection, due to microvascular dysfunction, when other routine vital parameters are still within normal ranges.

Objectives

Primary aim To assess, if pFTOE measured by five short NIRS (re-)applications within the first 6 hours after birth differs in neonates with early onset infection and neonates without infection.

Secondary aims To assess, if cerebral fractional tissue oxygen extraction (cFTOE) and cFTOE/pFTOE measured by five short NIRS (re-)applications within the first 6 hours after birth differs in neonates with early onset infection and neonates without infection. To assess, if there is a difference in pFTOE, cFTOE and cFTOE/pFTOE between term and preterm neonates.

Methods

Study population: Term and preterm neonates ≥30+0 weeks of gestation with respiratory distress and risk factors for infection admitted to the neonatal intensive care unit (NICU) on the first day after vaginal delivery or caesarean section on the first day after birth will be eligible for this study. Inclusion criteria are signs of respiratory distress at time-point of inclusion, age <6h and decision to conduct full life support. There will be four groups consisted with term(1) and preterm(2) neonates with early onset infection and term(3) and preterm(4) neonates without.

Procedure: Patients and maternal medical history, routinely sampled laboratory results and blood culture will be documented in each neonate.

Measurement: The NIRS-measurement will take place once within 6 hours after birth. For NIRS measurements the NIRO 200NX will be used and the NIRS sensors will be applied by hand on the right forearm (pTOI) and on the left forehead (cTOI) until stable signals are obtained for approximately 30 seconds, respectively. Then the sensors will be removed for 10sec rest period. After that the sensors will be reapplied in approximately the same positions. This procedure will be repeated five times.

Level of originality As many term and preterm neonates are admitted to the NICU after birth due to respiratory distress, there is growing interest in methods enabling to recognize subtle early signs like micro-vascular dysfunction due to infection. In the present study the investigators want to evaluate in neonates with respiratory distress if peripheral muscle and cerebral FTOE measured by short reapplications with NIRS in the first hours after birth enables to recognize early microvascular dysfunction and compromised oxygenation due to infections.

ELIGIBILITY:
Inclusion Criteria:

* Signs of respiratory distress at time-point of inclusion (tachypnoea >60/minutes, grunting, intercostal/subcostal/jugular retractions, nasal flaring, supplemental oxygen or respiratory upport)
* Decision to conduct full life support
* Written informed consent
* Age < 6 hours

Exclusion Criteria:

* No decision to conduct full life support
* no written informed consent
* gestational age <30+0 weeks of gestation
* age > 6 hours
* severe congenital malformations, severe asphyxia (umbilical cord artery pH <7.00)

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Term and preterm neonates ≥30+0 weeks of gestation with respiratory distress and risk factors for infection admitted to the Division of Neonatology, Department of Pediatrics and Adolescent Medicine, Medical University of Graz after vaginal delivery or caesarean section on the first day after birth will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-02-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
pFTOE | 5 minutes (duration of 5 re-applications)
  pFTOE within 6 hours after birth

SECONDARY OUTCOMES:
cFTOE | 5 minutes (duration of 5 re-applications)
  cFTOE and cFTOE/pFTOE within 6 hours after birth
gestational age | up to 10 weeks (until term age - discharge)
  term and preterm neonates

OTHER OUTCOMES:
TOI | 5 minutes (duration of 5 re-applications)
  cTOI, pTOI
routine monitoring data - arterial oxygen saturation (SpO2) | up to 10 weeks (until term age - discharge)
  SpO2 in percentage (%)
routine monitoring data - heart rate (HR) | up to 10 weeks (until term age - discharge)
  HR im beats per minute (bpm)
routine monitoring data - blood pressure (RR) | up to 10 weeks (until term age - discharge)
  RR in mmHg
routine monitoring data (temperature) | up to 10 weeks (until term age - discharge)
  temperature in °C
Laboratory parameter | up to 10 weeks (until term age - discharge)
  C reactive protein (mg/l) - routinely sampled
Laboratory parameter | up to 10 weeks (until term age - discharge)
  leukocytes (per µl) - routinely sampled
Laboratory parameter | up to 10 weeks (until term age - discharge)
  IT-ratio - routinely sampled
Laboratory parameter | up to 10 weeks (until term age - discharge)
  blood cultures - routinely sampled
Demographic data of the neonate | up to 10 weeks (until term age - discharge)
  gestational age (weeks)
Demographic data of the neonate | up to 10 weeks (until term age - discharge)
  birth weight (grams)
Demographic data of the neonate | up to 10 weeks (until term age - discharge)
  risk factors
Data of the neonate | up to 10 weeks (until term age - discharge)
  diagnosis (descriptive)
Data of the neonate | up to 10 weeks (until term age - discharge)
  therapy (descriptive)
Medication | up to 10 weeks (until term age - discharge)
  medication in appropriate dosage

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Pichler, Prof., MD, Principal Investigator — Medical University of Graz, Department of Pediatric and Adolescent Medicine, Division of Neonatology
Locations (1):
- Department of Pediatrics, Division of Neonatology, Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No